CLINICAL TRIAL: NCT05590559
Title: Ultrasound-guided Erector Spinae Plane Block Versus Paravertebral Block in Breast Cancer Patients Undergoing Mastectomy With Immediate Reconstruction - a Non-inferiority Trial. A Single-centre Randomized Controlled Non-inferiority Trial With a Parallel Group Design
Brief Title: Ultrasound-guided Erector Spinae Plane Block Versus Paravertebral Block in Breast Cancer Patients Undergoing Mastectomy With Immediate Reconstruction - a Non-inferiority Trial
Acronym: ESP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N20ESP
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer Patients Undergoing Mastectomy With Immediate Reconstruction
Keywords: Ultrasound-guided erector spinae plane block; paravertebral block
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paravertebral block (Active Comparator)
  Interventions: Drug: Morphine
- Ultrasound-guided erector spinae plane block (Experimental)
  Interventions: Other: Ultrasound-guided erector spinae plane block

INTERVENTIONS:
Drug: Morphine — Opiates
  Arms: paravertebral block
Other: Ultrasound-guided erector spinae plane block — PVB
  Arms: Ultrasound-guided erector spinae plane block

SUMMARY:
The objective of this study is to assess the non-inferiority of analgesic efficacy of ESP vs PVB for patients undergoing unilateral mastectomy followed by immediate reconstruction.

DETAILED DESCRIPTION:
n breast cancer treatment, surgery plays a central role in combination with chemotherapy, radiation and immunotherapy. Surgery may vary from conservative breast sparing interventions to large radical mastectomies with axillary lymph node dissection that require reconstructive (prosthetic) surgery. In many instances, reconstruction is not performed immediately, but immediate reconstruction is possible and offers many advantages to patients.

The Antoni van Leeuwenhoek hospital performs a large proportion (77%) of mastectomies with immediate reconstruction in the Netherlands. The combination of mastectomy with immediate reconstruction in one operation offers an extra challenge with regards to pain control. Post-operative pain is often treated with opioids, which has systemic side effects (nausea and vomiting). Opioids also inhibit cell-mediated immunity, which is a principal defense against cancer. Regional anesthetic techniques are often performed to reduce opioid consumption and enhance postoperative recovery. The current standard for regional anesthesia for breast surgery is the paravertebral block (PVB). This technique has the potential for severe complications such as epidural hematoma, hemo- or pneumothorax. The erector spinae plane block (ESP) was first described in 2016 as a novel regional anesthetic technique for acute and chronic thoracic pain. The site of injection is distant from the pleura, major blood vessels, and spinal cord; hence, the ESP block has relatively few contraindications and has therefore been suggested as an alternative to PVB when contra-indications, such as a bleeding diathesis, are present.Multiple studies have shown a decrease in opioid consumption in patients undergoing mastectomy, when ESP was compared to placebo. ESP has also been shown to be non-inferior to PVB for pain relief in patients undergoing thoracotomy. To date, only two studies have compared ESP to PVB for breast surgery, with conflicting results. In this study, we would like to investigate whether ESP can be considered non-inferior to PVB with regards to pain relief and use of opioids.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or older)
* ASA I-III
* Patients scheduled for elective unilateral mastectomy followed by direct reconstruction
* Ability to give written and oral informed consent

Exclusion Criteria:

* Patient refusal
* Non-elective surgery
* Any contraindication to paravertebral block (including bleeding diathesis, coagulopathy, severe pulmonary disease )
* Allergy to amide-linked local anesthetics
* Cardiac conductivity disorders (e:g: 2nd and 3rd AV-block)
* Severe spinal malformations or history of extensive spine surgery - A history of spinal cord injury
* Known psychiatric disorder
* Chronic pain patients or patients already using opioids pre-operatively
* Infection of the skin at the site of needle puncture area - Inability to give oral and written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult female patients
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference of highest numerical rating score (NRS - a linear 11 point scale for self-reported pain) during admission in the recovery room | 1 day
Difference in the ratio of the means of cumulative opioid dose (administered during admission in the recovery room) | 1 day

SECONDARY OUTCOMES:
Success rate as defined by satisfactory spread of local anaesthetic agents on ultrasound | 1 month
Ease of procedure (self-reported by anaesthetist on scale of 1-5) | 1 month
Total opioid dose administered on day 0 and on day 1 (iv, subcutaneous or oral - converted to morphine equivalent dose (MEQ) | 1 day after dose administration
Highest pain score on day 0 and 1 | 1 day
Time to readiness for discharge from the recovery room | 1 day
Complications of block (such as block failure, epidural hematoma, hemo- or pneumothorax and symptoms of toxicity of local anesthetics) | 1 day
Patient satisfaction on a scale of 0 (extremely unsatisfied) tot 10 (extremely satisfied) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- NKI-AvL, Amsterdam, North Holland, Netherlands